CLINICAL TRIAL: NCT03132870
Title: Predictive Diagnostic Criteria for Diagnosis of Transbronchial Biopsies, Echo-guided by Mini-probe in Peripheral Lung Lesions
Acronym: EBUS-R-PTB
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2016-40 Dr Basille
Record Dates: First submitted 2017-04-14; First posted 2017-04-28 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Transbronchial Biopsies; Peripheral Lung Lesion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Define predictive criteria for the diagnostic performance of echo-guide samples by mini-probe in peripheral lung lesions — Define predictive criteria for the diagnostic performance of echo-guide samples by mini-probe in peripheral lung lesions

SUMMARY:
The diagnosis of nodules and peripheral lung masses (lesions not accessible in classical bronchial endoscopy) is a challenge for the pulmonologist especially when these lesions are not accessible to the transparietal aspirate under scanner. The overall sensitivity of flexible fibroscopy for peripheral lesions is 69% (bronchial brushing, transbronchial biopsies, bronchoalveolar lavage and blind trans-mucosal aspiration). This sensitivity varies from 33% when the lesion is less than 2 cm, to 62% when it is greater than 2 cm. The puncture under scan of these lesions remains the gold standard. In the meta-analysis of Schreiber G et al., The diagnostic sensitivity of transparietal aspirate for peripheral lung lesions is 90%. On the other hand, the complication rate of this technique is not negligible, with in the study of Boskovic et al, a pneumothorax rate varying from 8 to 64%. In the literature, the only risk factor actually found is the existence of emphysema. However, thoracic drainage is rarely necessary.

Bronchial echo-endoscopy using a radial mini-probe was developed in 1992 by Thomas Hürter and Peter Hanrath to produce ultrasound guided specimens of these peripheral lung lesions. In the meta-analysis of Steinfort et al., The overall sensitivity of this mini-probe technique is 73% for the histological diagnosis. From the same author, a randomized trial compared the diagnostic sensitivity of transparietal aspirate undergoing ultrasound-guided transbronchial biopsy with a radial mini-probe: this was 93.3% versus 87.5% with no significant difference (p = 1 ), Whereas post-procedure complications are less frequent in the ultrasound procedure (27% versus 3%, p = 0.03). Steinfort also showed that the economic cost of bronchial echo-endoscopy by radial mini-probe and transthoracic puncture under CT was similar both to the success or failure of the first procedure requiring further investigations . Mini-probe-guided specimens are therefore an efficient diagnostic alternative to obtain a histological diagnosis of these peripheral lung lesions

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent mini-probe fibroscopy at Amiens University Hospital from January 2013 to March 2016

Exclusion Criteria:

* No

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a mini-probe fibroscopy
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Analyze predictive criteria of the performance diagnosis by echo-guide sampling by mini-probe | 39 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France